CLINICAL TRIAL: NCT04879693
Title: Effectiveness and Safety of the Dexcom G6 Continuous Glucose Monitoring System in Non-Critically Ill Patients in the Inpatient Setting
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: DexCom, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PTL-904283
Record Dates: First submitted 2021-05-05; First posted 2021-05-10 (Actual); Last update posted 2021-05-10 (Actual); Status verified 2021-05

CONDITIONS: Patients Needing Glucose Control
MeSH Terms: interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Masking Description: All systems worn will be blinded. All sensor insertions will be performed at the clinic by subjects and/or caregivers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Hospitalized Patients (Experimental): To assess performance of CGM compared to comparator measurement.
  Interventions: Device: Continuous Glucose Monitoring System

INTERVENTIONS:
Device: Continuous Glucose Monitoring System — Continuous Glucose Monitoring System

SUMMARY:
Effectiveness and Safety of the Dexcom G6 Continuous Glucose Monitoring System in Non-Critically Ill Patients in the Inpatient Setting

DETAILED DESCRIPTION:
To assess the performance of the CGM System in comparison to a blood glucose comparator method in non-critically ill hospitalized patients who need glucose control.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older
* Admitted to the hospital in a non-ICU bed or once transferred out of ICU
* Anticipate at least 48 hours of hospital stay
* On treatment for glucose control.
* Willingness to complete the study.
* Willingness to wear up to 3 CGM systems simultaneously. Two in the abdomen and one on the back of the arm or one on each arm and one on the abdomen.
* Subject and/or caretaker are able to speak, read, and write English

Exclusion Criteria:

* Presence of extensive skin changes/diseases at sensor wear site(s) that preclude wearing the sensor(s) on normal skin (e.g., extensive psoriasis, recent burns or severe sunburn, extensive eczema, extensive scarring, extensive tattoos, dermatitis herpetiformis)
* Currently in an intensive care unit (ICU) of the following type (does not apply to participants placed in an ICU bed due to space issues in the non-ICU areas)
* Known allergy to medical-grade adhesives
* Pregnancy, demonstrated by a positive test (for subjects of childbearing potential)
* Women admitted to give birth or any other admission related to pregnancy
* Patients receiving Hydroxyurea
* Bleeding disorder
* Participants that are currently being treated for malignancies, cancer
* Participant that are hospitalized to receive an organ transplant
* Require a Magnetic Resonance Imaging (MRI) scan
* End stage renal disease and currently managed by dialysis or anticipating initiating dialysis during the study wear period
* Current participation in another investigational study protocol (If a subject has recently completed participation in another drug study, the subject must have completed that study at least 7 days prior to being enrolled in this study.)
* Any condition that, in the opinion of the Investigator, would interfere with their participation in the trial or pose an excessive risk to study staff (e.g., known history of hepatitis B or C)

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2021-06 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
System Performance | Up to 10 days
  Assess the performance of the CGM System in comparison to a blood glucose comparator method in non-critically ill hospitalized patients who need glucose control.

IPD SHARING:
Plan to Share IPD: No